CLINICAL TRIAL: NCT04819529
Title: Early and Intensive Occupational Therapy Improves the Functional Status of Critical Patients Undergoing Mechanical Ventilation at Discharge: Randomized Clinical Trial
Brief Title: Early and Intensive Occupational Therapy in Mechanical Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Hospital Base Valdivia (Unknown); Hospital Santiago Oriente - Dr. Luis Tisné Brousse (Unknown)
Responsible Party: Principal Investigator, Eduardo Tobar, Associated professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA19I0138
Record Dates: First submitted 2021-03-03; First posted 2021-03-29 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Critical Illness; Ventilator Lung; Impairment, Cognitive; Impairment, Coordination
MeSH Terms: conditions — Critical Illness; Cognitive Dysfunction; Ataxia

STUDY DESIGN:
Intervention Model Description: A control group (standard ASDM measures) or an intervention group (early and intensive occupational therapy + ASDM) will be randomized. The intervention group will receive 20 occupational therapy sessions. The interventions will be organized on the basis of i) level of sedation, ii) presence or absence of delirium (according to CAM ICU +/- (Confusion Assessment Method Intensive Care Unit)), iii) movement with or without gravity (cut-off point 3 points in elbow flexion movement in Medical Research Council(MRC)). The areas of intervention implemented by occupational therapist will be: i) Polysensory stimulation, ii) Cognitive stimulation, iii) Basic activities of daily living, iv) Motor function stimulation, v) Education
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, researchers, recruiters, evaluators, control group team and data analyst will be masked. These teams will not have contact with the interventionists of the experimental group. Evaluators who have contact with the patients of both groups, they will be professionals from other medical units, who do not know the ICU team, and will only be able to maintain their dialog, according to the guideline of each evaluation.
  It is not possible to mask the treating occupational therapist and patient receiving OT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Early and intensive Occupational Therapy (Experimental): These sessions will be implemented by occupational therapists trained in ICU, who will conduct 20 sessions of 30 min, distributed depending on the level of sedation, i) SAS (Sedation-Agitation Scale) 1 patients have one session each 48 h, evaluating the change of sedation level each 24 h; ii) SAS 2 patients have one session each 24 h, iii) SAS 3-5 have two sessions every day. The sessions will begin once the patient needs mechanical ventilation for at least 12 h
  Interventions: Behavioral: Early and Intensive Occupational Therapy
- Control group - Standard Analgesia,Sedation, Delirium and Mobilization (ASDM) Protocol (No Intervention): The ASDM protocol will be implemented to mechanically ventilated patients in the ICU, following the aspects recommended by experts and the current evidence. For this, the team of medical, nurses, and physiotherapist will be trained to understand and facilitate the ASDM actions that each one must implement.

INTERVENTIONS:
Behavioral: Early and Intensive Occupational Therapy — Occupational therapists will implement the following activities:
  * Polysensory stimulation: external stimulation for increasing the level of alertness. It will be implemented with SAS 1 one session each 48 h and SAS 2 one session each 24 h.
  * Cognitive stimulation: bundle of exercises for activating mental functions, i.e: alertness, visual perception, memory, calculus, problem solving, praxis, language. Patients with SAS 3, 4 and 5. In SAS <2, 6> environmental orientation will be considered
  * Basic activities of daily living (BADLs): promotion of independence that initially practice hygiene, personal grooming. Patients with SAS 3, 4 and 5
  * Motor function Stimulation: exercises to keep the patient's upper extremities active and functional. Patients with SAS with 3,4 and 5. Patients with SAS 1 and 2 will use adaptations to prevent edema and bedsores on vulnerable body areas
  * Education: daily visits by trained family members and health staff about the intervention process
  Arms: Experimental Group - Early and intensive Occupational Therapy

SUMMARY:
This study evaluates the efficacy of an early and intensive occupational therapy (OT) protocol in critical adult patients requiring mechanical ventilation. Evaluating the functional independence at hospital discharge.

DETAILED DESCRIPTION:
A randomized clinical trial with an experimental-control will be implemented, considering the prospective multicenter group, with parallel groups, in a 1:1 ratio, in 3 Chilean hospitals.

A control group will has a standard analgesia, sedation, delirium and mobilization (ASDM) measures or an intervention group will have early and intensive OT plus ASDM.

The intervention group will receive 20 OT sessions, mainly twice a day, which considers a predefined protocol of actions according to the patient's condition

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years.
* Need for hospitalization in ICU.
* At least 12 h of invasive mechanical ventilation
* Informed consent signed by legal representative and / or patient.

Exclusion Criteria:

* Known cognitive impairment before admission with short IQCODE (Informant Questionnaire on Cognitive Decline in the Elderly) Scores> 3.3 were excluded.
* Previous functional impairment, FAQ (Functional Activities Questionnaire) defined as > 6 points.
* Severe communication disorder and cultural limitation of language (language different from Spanish)
* Patient with limited therapeutic proportionality.
* Neurocritical patients (moderate-severe Traumatic Brain Injury / stroke of some kind / among others)
* Spinal injury or unstable fractures that limit mobilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional independence at hospital discharge | Day 28 (+/- 3 days) from beginning of mechanical ventilation
  The FIM (Functional independence measure) instrument will be applied by evaluator team. This scale shows that higher score is better, which will be compared between control and experimental group

SECONDARY OUTCOMES:
Delirium-free days | Defined as the number of days in the first 14 days with the CAM-ICU instrument negative and non-coma day.
  CAM-ICU (Confusion Assessment Method Intensive Care Unit) instrument will be applied once a day by evaluator
Coma-free days | Defined as the number of days in the first 14 days with the SAS.
  SAS (Sedation-Agitation Scale) instrument will be applied once a day by evaluator. If SAS 1-2: coma day
Delirium-coma free days | Defined as the number of days in the first 14 days with the SAS and CAM-ICU
  SAS and CAM-ICU instruments will be applied once a day by evaluator. Every day without coma or delirium its an delirium-coma free day
Hazard ratio for delirium in the interventional versus control group | Collecting from the first 14 days with the CAM-ICU instrument and coma.
  A composite analysis who involves delirium-coma free days to day 14. Hazard Ratio <1 interpreted as a lower daily hazard of delirium - implying a shorter mean duration of delirium among days at risk for delirium
Cognitive status of patients | Day 28 (+/- 3 days) from beginning of mechanical ventilation and day 90 (+/- 7 days)after hospital discharge
  MoCA (Montreal Cognitive Assessment) instrument (cognitive status).This scale shows that higher score is better, which will be compared between control and experimental group
Motor status of patients | Day 28 (+/- 3 days) from beginning of mechanical ventilation
  Grip strength (motor status) with dynamometer will be applied by evaluator. This scale shows that higher score is better, which will be compared between control and experimental group
Quality of life of patients | Day 90 (+/- 7 days) from beginning of mechanical ventilation
  EQ-5D-5L (Euro Qol 5 dimensions 5 level) will be applied by evaluator. It will be considered a cut-off point in the Chilean population
Mental health | Day 90 (+/- 7 days) from beginning of mechanical ventilation
  Hospital Anxiety and Depression Scale (HADS) will be applied by evaluator. This scale shows that lower score is better, which will be compared between control and experimental group
Functional independence | Day 90 (+/- 7 days) from beginning of mechanical ventilation
  The FIM (Functional independence measure) instrument will be applied by evaluator. This scale shows that higher score is better, which will be compared between control and experimental group

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmerman JE, Kramer AA, Knaus WA. Changes in hospital mortality for United States intensive care unit admissions from 1988 to 2012. Crit Care. 2013 Apr 27;17(2):R81. doi: 10.1186/cc12695. PMID 23622086
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] van der Schaaf M, Beelen A, Dongelmans DA, Vroom MB, Nollet F. Functional status after intensive care: a challenge for rehabilitation professionals to improve outcome. J Rehabil Med. 2009 Apr;41(5):360-6. doi: 10.2340/16501977-0333. PMID 19363570
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Marra A, Ely EW, Pandharipande PP, Patel MB. The ABCDEF Bundle in Critical Care. Crit Care Clin. 2017 Apr;33(2):225-243. doi: 10.1016/j.ccc.2016.12.005. PMID 28284292
- [Background] Costigan FA, Duffett M, Harris JE, Baptiste S, Kho ME. Occupational Therapy in the ICU: A Scoping Review of 221 Documents. Crit Care Med. 2019 Dec;47(12):e1014-e1021. doi: 10.1097/CCM.0000000000003999. PMID 31738741
- [Result] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Result] Sacanella E, Perez-Castejon JM, Nicolas JM, Masanes F, Navarro M, Castro P, Lopez-Soto A. Functional status and quality of life 12 months after discharge from a medical ICU in healthy elderly patients: a prospective observational study. Crit Care. 2011;15(2):R105. doi: 10.1186/cc10121. Epub 2011 Mar 28. PMID 21443796
- [Result] Alvarez EA, Garrido MA, Tobar EA, Prieto SA, Vergara SO, Briceno CD, Gonzalez FJ. Occupational therapy for delirium management in elderly patients without mechanical ventilation in an intensive care unit: A pilot randomized clinical trial. J Crit Care. 2017 Feb;37:85-90. doi: 10.1016/j.jcrc.2016.09.002. Epub 2016 Sep 10. PMID 27660922
- [Derived] Alvarez E, Garrido M, Salech F, Rojas V, Jara N, Farias JI, Ponce D, Tobar E. Early occupational therapy in mechanically ventilated patients improves functional status: Study protocol. Br J Occup Ther. 2023 Nov;86(11):728-739. doi: 10.1177/03080226231184992. Epub 2023 Jul 14. PMID 40336796